CLINICAL TRIAL: NCT06911294
Title: Feasibility of InnovaTive Approaches for Personalized Cardiovascular PREVention: Randomized Controlled Pilot Trial and Multidisciplinary Evaluation for National Health Service Implementation
Brief Title: Feasibility of Innovative Approaches for Personalized Cardiovascular Prevention
Acronym: FITPREV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Roberta Pastorino, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7700, 7885-7890
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: Coronary Heart Disease
Keywords: coronary artery disease; Polygenic Risk Score
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Genetic Risk Score | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No intervention - Standard of Care (No Intervention): Participants will receive traditional lifestyle advices in order to reduce the risk.
- Genetic testing - PRS (Experimental): Arm Description: Participants will receive the information of the genetic cardiovascular risk (PRS) and personalized advices.
  Interventions: Behavioral: Polygenic Risk Score
- Experimental: Digital intervention - app and wearable device (Experimental): Arm Description: Participants will receive an app and a wearable device for the evaluation of various parameters.
  Interventions: Behavioral: Digital app and wearable device
- Digital intervention and genetic testing - PRS (Experimental): Arm Description: Participants will receive both app and wearable device and PRS information
  Interventions: Behavioral: Polygenic Risk Score; Behavioral: Digital app and wearable device

INTERVENTIONS:
Behavioral: Polygenic Risk Score — genetic test for the evaluation of cardiovascular risk
  Arms: Digital intervention and genetic testing - PRS; Genetic testing - PRS
Behavioral: Digital app and wearable device — a wearable device connected with its app
  Arms: Digital intervention and genetic testing - PRS; Experimental: Digital intervention - app and wearable device

SUMMARY:
The goal of the FITPREV (Feasibility of InnovaTive approaches for personalized cardiovascular PREVention: randomized controlled pilot trial and multidisciplinary evaluation for National Health Service implementation) clinical trial is to study the feasibility of innovative approaches( Polygenic Risk Score and health smartwatch) for personalized primary preventive interventions in cardiovascular diseases (CVD). The main questions it aims to answer are:

* Feasibility of a greater study.
* Feasibility of the interventions in a realistic setting, such as the medical office of a General Practitioner.

Participants will be randomized in one of the four parallel arms:

* standard of care;
* genetic testing for cardiovascular genetic risk (through the cardiovascular Polygenic Risk Score or PRS);
* digital intervention with a wearable device and its app;
* digital intervention and genetic testing

The primary outcomes that are going to be evaluated are patient's and General Practitioners' overall judgment of the study and its feasibility.

Secondarily the efficacy of returning Polygenic Risk Score (PRS) results will be assessed. This will happen on two endpoints: i) change in lifestyle pattern; ii) CVD risk profile modification. The postulated hypothesis is that the achievement of these endpoints is more likely in presence of at least one of the aforementioned interventions than among subjects who receive only traditional risk assessment at baseline.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility and secondarily efficacy of disclosing cardiovascular genetic risk-in the setting of a general practitioner's office-in the promotion of healthier lifestyle behaviors.

The enrollment period will last 6 months, with each participant taking part in the study for 12. There are three key time points in the study, T0 or baseline (enrollment phase), T1 or disclosure visit after one month, T2 intermediate visit(after six months) and T3 or final visit at 12 months. At enrollment, participants will be classified into risk categories based on cardiovascular risk using the SCORE-2 or SCORE 2-OP tool. Individuals aged 40-69, without diabetes or congenital hypercolesterolemia, with a SCORE-2 between 2.5% and 10% and a diagnosys of metabolic syndrome according to the American Hearth Association Criteria will be enrolled.

Once enrolled (T0), all participants will sign the informed consent form and undergo a comprehensive assessment, which includes:

* Completing a questionnaire on socioeconomic status, area of residence, and lifestyle, using the Life's Essential 8 tool. The questionnaire will cover smoking status, alcohol consumption, dietary pattern, sleep pattern, and physical activity. Participants will be classified into favorable, intermediate, or unfavorable individual lifestyle patterns according to the Life's Essential 8 score.
* Blood analysis will be performed to evaluate the lipid profile, including total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides.

At T1, a disclosure visit will be conducted to explain the assigned lifestyle category, share the results of the blood tests, and provide information on the expected interventions based on the assigned group.

The questionnaire will be administered at T0, T2, and T3. Blood analysis and cardiovascular profile evaluation will be conducted at both T0 and T3.

Feasibility Questionnaire: Both participants and medical professionals will complete a questionnaire on the acceptability and feasibility of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-69 years;
* 10 year cardiovascular risk score SCORE2 between 2.5% and 10%.
* Diagnosis of metabolic syndrome according to the American Heart Association criteria , defined as the presence of three or more of the following:

  * Central or abdominal obesity, measured by waist circumference (greater than 40 inches - 102 cm in men and 35 inches - 89 cm in women).
  * Elevated triglycerides: levels equal to or greater than 150 mg/dL or use of medication for hypertriglyceridemia.
  * Low HDL cholesterol levels (less than 40 mg/dL in men and less than 50 mg/dL in women) or use of cholesterol-lowering medication.
  * Elevated blood pressure: systolic ≥130 mmHg or diastolic ≥85 mmHg, or use of antihypertensive medication.
  * Elevated fasting blood glucose: ≥100 mg/dL or use of glucose-lowering medication.

Exclusion Criteria:

* Diabetes:
* Familial hypercholesterolemia;
* Previous cardiovascular events.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility for the patients | 1 year
  Feasibility will be measured scoring the answer to a short questionnaire compiled at the end of the study(Using one open question, a few yes/no questions and some questions with a Likert 5 scale of agreement).
Feasibility for the General Practitioners | 1 year
  Feasibility will be measured scoring the answer to a short questionnaire compiled at the end of the study(Using one open question, a few yes/no questions and some questions with a Likert 5 scale of agreement).

SECONDARY OUTCOMES:
Change in the Lifestyle Category | 12 months
  The lifestyle category will be measured using the Life's Essential 8 tool. A change will be considered achieved if there is a shift towards a more favorable lifestyle category.
Modification of the Lipid Profile | 12 months
  We will evaluate whether there is a change in the lipid profile compared to the baseline value. The modification of the lipid profile can also be considered as an indicator of the modification of the cardiovascular risk profile measured with the SCORE 2 charts.

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - Studio Antonaci, Rome, Italy
  - Studio Colletti, Rome
  - Studio Maggiori, Rome
  - Studio Mammucari, Rome
  - Studio Marra, Rome
  - Studio Paoletti, Rome
  - Studio Pasca, Rome

REFERENCES:
- [Background] Lloyd-Jones DM, Allen NB, Anderson CAM, Black T, Brewer LC, Foraker RE, Grandner MA, Lavretsky H, Perak AM, Sharma G, Rosamond W; American Heart Association. Life's Essential 8: Updating and Enhancing the American Heart Association's Construct of Cardiovascular Health: A Presidential Advisory From the American Heart Association. Circulation. 2022 Aug 2;146(5):e18-e43. doi: 10.1161/CIR.0000000000001078. Epub 2022 Jun 29. PMID 35766027